CLINICAL TRIAL: NCT06855563
Title: Cities for Better Health Childhood Obesity Prevention Initiative: A Multi-country Community-based Prevention and Intervention Project Targeting Childhood Obesity Through Diet and Physical Activity Interventions in Disadvantaged Communities of Urban Areas
Brief Title: Cities for Better Health Childhood Obesity Prevention Initiative
Acronym: CBH COPI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAS-8381; U1111-1314-3391 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention packages are expected to consist of multiple specific activities tailored to the local context. All intervention packages will be designed to be (i) multi-level (i.e. targeting at least two of individual, external and structural environments), (ii) multi-component (i.e. targeting both healthy diet and physical activity), (iii) co-created with local communities in which they are implemented and (iv) health equity oriented in terms of both access and improvement. The exact package of interventions will differ by country and is expected to evolve pragmatically over time.
  The intervention group in each country will be made up of (children in) neighbourhoods where intervention packages are implemented.
  Interventions: Behavioral: Community-based intervention packages
- Comparison group (No Intervention): The comparison group will be made up of (children in) neighbourhoods where intervention packages are not implemented.

INTERVENTIONS:
Behavioral: Community-based intervention packages — Community-based intervention packages
  * Intervention packages are expected to consist of multiple specific activities tailored to the local context. All intervention packages will be designed to be (i) multi-level (i.e. targeting at least two of individual, external and structural environments), (ii) multi-component (i.e. targeting both healthy diet and physical activity), (iii) co-created with local communities in which they are implemented and (iv) health equity oriented in terms of both access and improvement. The exact package of interventions will differ by country and is expected to evolve pragmatically over time.
  * The intervention group in each country will be made up of (children in) neighbourhoods where intervention packages are implemented.
  Arms: Intervention group

SUMMARY:
This research project is part of the 'Cities for Better Health Childhood Obesity Prevention Initiative' (CBH COPI). The objective of the CBH COPI initiative is to develop, implement, and evaluate the effectiveness of a package of prevention interventions in five cities to promote healthy eating, physical activity, a positive health-related quality of life, and a reduction in rates living with overweight or obesity among children aged 6-13 years in six cities across Australia, Brazil, Canada, Japan, South Africa and Spain.

The primary research objective of CBH COPI is to estimate the impact of the intervention packages on the average BMI of the target population of children across the participating countries, at one-year and two-year follow-ups. The secondary research objective is to estimate the impact of the intervention packages on average health-related quality of life (HRQoL) at the same time points. Exploratory aims include estimating the impact of the packages on behaviours related to physical activity and diet.

DETAILED DESCRIPTION:
Requirements for interventions:

The interventions in each country will be multi-level multi-component (MLMC) community-based packages. Their exact features will be tailored to the needs and opportunities of each participating country.

Requirements for study design:

The minimum evaluation study design in terms of robustness is a repeated cross-sectional study with a comparison group. This involves measuring outcomes in a cross-section of children living in the intervention areas of a participating city (i.e. the areas in which the CBH COPI interventions were implemented) and a cross-section of children in similar comparison areas in which the interventions were not implemented, before and after the interventions are introduced. The global analysis will then compare trends in outcomes between intervention- and comparison-group areas. Countries are allowed to implement more robust designs (e.g. incorporating randomisation) if this is feasible.

Each country-level study will collect a set of prespecified indicators at baseline and at two subsequent follow-ups (after 10-12 months, and after 20-24 months). The primary outcome indicator is BMI z-score and the required secondary and exploratory outcomes are defined above. A list of sociodemographic indicators (age, sex, ethnicity, household affluence) is also required to be collected (unless this is not feasible in an individual country for legal reasons).

It is anticipated that 2,000 children in the target population will be recruited per data collection point (baseline, first follow-up, second follow-up) in each country. It is recommended (as the default option) that data are collected from 20 'clusters' (schools) from at least 10 'neighbourhoods' (administrative areas or school catchment areas, depending on the country) over these time points. This set up gives a minimum detectable effect size of Cohen's d = 0.15 in country-level analyses. The sample of neighbourhoods/clusters will be chosen according to feasibility and representativeness considerations in each country.

Local evaluations will be adapted to fit with the social, cultural and policy landscape of each implementing site.

ELIGIBILITY:
To be eligible to be involved in data collection, children must attend the 'clusters' (schools) that are part of the study. In each cluster, country evaluation teams will try to ensure that the sample of children selected for data collection is representative of the total population in that cluster (e.g. the full list of students ages 6-13 who go to that school) - in particular, with respect to age and sex.

All countries will also use the inclusion and exclusion criteria below for children in the study:

Inclusion Criteria:

* Informed consent obtained by the child's parent or legal guardian before any study-related activities (where study-related activities are defined as any procedure related to recording of data according to the protocol). The specific consent form and procedures for obtaining consent will be outlined by the local project partner.
* Aged 6-13 years (both 6 and 13 allowed) at the time of signing consent. Deviations from or exceptions to this procedure must be agreed between the research team in the relevant country and the GIP, and are subject to the relevant local ethical amendment procedure. The exception must be due to a scientifically sound rationale and must further consider the following guiding principles: "it must be measurable, it must have marginal utility, it must be meaningful (i.e. linked to the ultimate impact and the primary and/or secondary objective)".

Exclusion Criteria:

- Children will be excluded from the study if their parent(s) do not provide fully informed consent for their data to be collected, if during the measurement day they do not agree to participate, or if the child's parent(s) or legal guardian(s) withdraw their consent for their child participating in the research at any point in line with processes described in local informed consent forms.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36000 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index z-score (BMI-z) adjusted for age and sex | At baseline, 1st follow-up (10-12 months) and 2nd follow-up (20-24 months)
  z-score

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL), proxied by KIDSCREEN-10 index | At baseline, 1st follow-up (10-12 months) and 2nd follow-up (20-24 months)
  Constructed from KIDSCREEN-10 survey. Each of the 10 measures is coded from 1-5. Sum across 10 measures to create a total score (10-50) and linearly rescale to 0-100 for interpretation.

OTHER OUTCOMES:
Physical activity outcomes | At baseline, 1st follow-up (10-12 months) and 2nd follow-up (20-24 months)
  Physical activity outcomes will be elicited via survey instruments adapted from the Core Indicators and Measures of Youth Health - Physical Activity & Sedentary Behavior Module questionnaire. The main physical activity outcomes are: MVPA time (mins per day), physical activity time (mins per day), sedentary time (mins per day), energy expended through physical activity (kcal per day).
Diet outcomes | At baseline, 1st follow-up (10-12 months) and 2nd follow-up (20-24 months)
  Diet outcomes will be measured with an edited version of the Diet Quality Questionnaire (DQQ). The main diet outcome is the Global Dietary Recommendations (GDR) score, and other outcomes include energy intake, nutritional intake and intake of specific food groups.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (6):
- Novo Nordisk Investigational Site, Loagan, Australia
- Novo Nordisk - Türkiye, Bangalore, Brazil
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk - Türkiye, Bangalore, Japan
- Novo Nordisk Investigational Site, Johannesburg, South Africa
- Novo Nordisk Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com